CLINICAL TRIAL: NCT05913648
Title: Urdu Translation, Validity and Reliability of Menopause-specific Quality of Life Scale
Brief Title: Urdu Version of Menopause-specific Quality of Life Scale
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: RiphahIU Khansa Ishaq
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Menopause

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tool Translation — The Data Collection procedure will be done in two phases. The first phase will revolve around the translation of the instrument. Firstly the tool will be translated into Urdu with the help of two professional translators and then it will be back-translated into English to cross-check the clarity of the text. The translation will focus more on the context and understanding of the text rather than literal word-to-word meanings. The translation will be done according to the WHO guidelines. The Urdu version of MENQOL will be used to assess content validity on menopausal women.

SUMMARY:
Menopause is accompanied by a spectrum of symptoms that are frequently related to hormonal changes. Menopause and its symptoms frequently have an impact on postmenopausal women's Quality of Life. There is a need for culturally adapted screening tool to aid healthcare professionals or clinicians to screen the symptoms of menopausal women, so the aim of this study is to translate the Menopause specific quality of life (MENQOL) into Urdu and to find the reliability and validity of the translated version Menopause specific quality of life in menopausal women.

DETAILED DESCRIPTION:
Menopause is accompanied by a variety of physiological changes and symptoms, including hot flashes, nightly sweating, anxiety, headaches, vaginal dryness, lethargy, irritability, and sleep disturbance. Menopause and its symptoms frequently have an impact on postmenopausal women's quality of life, a metric that is influenced by a variety of societal and personal circumstances. The Menopause-Specific Quality of Life Questionnaire(MENQOL) evaluates the prevalence and severity of bothersome physical and psychological concerns that women could experience during the menopausal transition.

As cross-border and cross-cultural studies continue to increase, there is a greater need for linguistic validation of tools in various societies. Until now no translation or adaptation of the MENQOL questionnaire has been made for the population with different languages in Pakistan. There is a need for culturally adapted screening tools to aid healthcare professionals or clinicians to screen the symptoms of menopausal women in the Pakistani population. As the Urdu language is Pakistan's national language so commonly used all over Pakistan, so it is required to translate and culturally adapt the MENQOL scale into Urdu language for the Pakistani population.

ELIGIBILITY:
Inclusion Criteria:

* Natural Menopause
* Females who are able to speak and read Urdu
* Volunteer to participate in the study

Exclusion Criteria:

* Mental in capacity to complete a self-administered questionnaire
* Communication problem
* Taking treatment for menopausal symptoms
* History of hysterectomy or ovariectomy
* Any systemic Chronic diseases affecting quality of life

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women after menopause will be recruited to report their quality of life domains on the translated version of MENQOL scale
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Menopause-specific quality of life (MENQOL) | Baseline
  The Menopause-Specific Quality of Life (MENQOL) questionnaire is a tool designed to assess the quality of life of women who are experiencing menopause. It consists of 29 items that measure the impact of menopausal symptoms on four domains: vasomotor (item 1-3). Psychological (items 4-10), physical (items 11-26) and sexual (items 27-29). The higher score indicates the symptom is more bothersome whereas the lower score indicates the symptoms are not at all bothered.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Ghosia medical center, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beura S, Patnaik L, Sahu M. Translation, Reliability, and Validity Test of Odia Version of Menopause-Specific Quality of Life Questionnaire Among Postmenopausal Women for Menopausal Symptoms. J Midlife Health. 2022 Apr-Jun;13(2):121-126. doi: 10.4103/jmh.jmh_222_21. Epub 2022 Sep 16. PMID 36276615
- [Background] Rathnayake N, Alwis G, Lenora J, Mampitiya I, Lekamwasam S. Linguistic and psychometric validation of sinhala version of menopause specific quality of life questionnaire. Sri Lanka J Soc Sci. 2021;44(1):15-26.
- [Background] Papadima EI, Boutsiadis A, Soldatou A, Ivanidou S, Vassilakou T, Michala L. Linguistic translation and validation of the Menopause-specific Quality of Life (MENQOL) questionnaire in Greek menopausal women. Menopause. 2020 Jul;27(7):808-815. doi: 10.1097/GME.0000000000001527. PMID 32217885
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630